CLINICAL TRIAL: NCT00692900
Title: Phase I Dose-Escalation Parallel Studies of Intraperitoneal Oxaliplatin With Intravenous Docetaxel and Intravenous Oxaliplatin With Intraperitoneal Docetaxel in Platinum-Sensitive or Platinum-Resistant Recurrent Ovarian, Primary Peritoneal, and Fallopian Tube Cancer
Brief Title: Safety Study Involving Oxaliplatin With Docetaxel for Recurrent Ovarian,Primary Peritoneal, and Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Robert Edwards, Principal Investigator, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OX-06-009
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): intravenous (IV) docetaxel and intraperitoneal (IP) oxaliplatin
  Interventions: Drug: intravenous docetaxel with intraperitoneal oxaliplatin
- 2 (Experimental): intravenous (IV) oxaliplatin and intraperitoneal(IP) docetaxel
  Interventions: Drug: intravenous oxaliplatin with intraperitoneal docetaxel

INTERVENTIONS:
Drug: intravenous docetaxel with intraperitoneal oxaliplatin — IV docetaxel 75 mg/m2 over 1 hour on day #1 followed by intraperitoneal oxaliplatin escalating from 50 mg/m2 on day #2. Cycles of treatment will be repeated every 3 weeks until disease progression or intolerable toxicity occurs.
  Arms: 1
Drug: intravenous oxaliplatin with intraperitoneal docetaxel — IV oxaliplatin 75 mg/m2 over 1 hour on day #1 followed by intraperitoneal docetaxel escalating from 50 mg/m2 on day #2. Cycles of treatment will be repeated every 3 weeks until disease progression or intolerable toxicity occurs.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safest and maximum tolerated dosing regimens for intraperitoneal oxaliplatin with intravenous docetaxel and intravenous oxaliplatin with intraperitoneal docetaxel for recurrent ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
This is a non-randomized, open-label Phase I trial in patients with previously treated, recurrent ovarian, primary peritoneal, or fallopian tube cancer. Patients may have either platinum -sensitive (relapse > 12 months from primary therapy) or platinum-resistant (relapse ≤ 12 months from primary therapy) disease.

Up to 20 patients will be enrolled into each of the following arms:

* Arm 1 patients will receive intravenous docetaxel at standard dosing of 75 mg/m2 over 1 hour on day #1 followed by intraperitoneal oxaliplatin on day #2 until maximum tolerated dose is achieved.
* Arm 2 patients will receive intravenous oxaliplatin at standard dosing of 75 mg/m2 over 1 hour on day #1 followed by intraperitoneal docetaxel on day #2 until maximum tolerated dose is achieved.

Treatment will be repeated every 3 weeks until disease progression, intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent histologically confirmed platinum-sensitive or platinum-resistant ovarian, primary peritoneal, or fallopian tube cancer
* Subjects may not have had > 3 prior regimens and must not have had a platinum or taxane agent within the past 6 months. Last chemotherapy must have been > 4 weeks prior to enrollment. Subjects may not have had prior whole abdomen or pelvic radiation. Patients may not have had > 6 cycles of an alkylating agent or > 450 mg/m2 of doxorubicin.
* ECOG Performance Score of ≤2 (Appendix A)
* Adequate bone marrow as evidenced by:

  * Absolute neutrophil count > or equal to 1,500/uL
  * Hemoglobin > or equal to 8 g/dl
  * Platelet count > or equal to 100,000/uL
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin < 1.5 mg/dL
  * Alk Phos, AST/ALT must be < 3x ULN or <5x ULN if hepatic mets.
  * AST/ALT < 3X the ULN for the reference lab
* Patients must be recovered from both the acute and late effects of any prior surgery, radiotherapy or other antineoplastic therapy
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

* Patients with an active infection or with a fever > 101.30 F within 3 days of the first scheduled day of protocol treatment
* Patients with active extra-abdominal metastases
* Patients with active CNS metastases. Patients with stable CNS disease, who have undergone radiotherapy at least 4 weeks prior to the planned first protocol treatment and who have been on a stable dose of corticosteroids for 3 weeks are eligible for the trial
* History of prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin or cervical intra-epithelial neoplasia
* Patients with known hypersensitivity to any of the components of docetaxel or oxaliplatin
* Patients who received pelvic or abdominal radiotherapy
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Peripheral neuropathy ≤ Grade 2
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of allogeneic transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the safest and maximum tolerated dose regimen for IV oxaliplatin with intraperitoneal docetaxel and IV oxaliplatin with intraperitoneal docetaxel in patients with recurrent ovarian, primary peritoneal, or fallopian tube cancer. | 18 months

SECONDARY OUTCOMES:
To assess quality of life | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Edwards, MD, Principal Investigator — University of Pittsburgh Medical Center; Kristin Zorn, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States